CLINICAL TRIAL: NCT02472704
Title: Lymphocytic Enteritis and Suspected Coeliac Disease: Double-blind Gluten vs Placebo Rechallenge
Brief Title: Lymphocytic Enteritis and Suspected Coeliac Disease: Gluten vs Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Principal Investigator, Fernando Fernandez-Bañares, Dr, Hospital Mutua de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSG-DC/01/01
Record Dates: First submitted 2015-06-09; First posted 2015-06-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Celiac Disease; Non-celiac Gluten Sensitivity
Keywords: celiac disease; lymphocytic enteritis; non-celiac gluten sensitivity; double-blind gluten rechallenge
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gluten challenge (Active Comparator): Gluten powder (10 g every 12 hours), 24 weeks
  Interventions: Dietary Supplement: Gluten challenge
- Placebo challenge (Placebo Comparator): Placebo (maltodextrin; 10 g every 12 hours), 24 weeks
  Interventions: Dietary Supplement: Placebo challenge

INTERVENTIONS:
Dietary Supplement: Gluten challenge — gluten (20 g/day) (identical powder sachets than placebo, mixed with meals) rechallenge while on a gluten-free diet
  Arms: Gluten challenge
Dietary Supplement: Placebo challenge — placebo (maltrodextrin) (identical powder sachets than gluten, mixed with meals) rechallenge while on a gluten-free diet
  Arms: Placebo challenge

SUMMARY:
Patients with lymphocytic enteritis (LE), HLA-DQ2/8+, negative celiac serology and clinical and histological response to a gluten-free diet (GFD) do not fulfil the diagnostic criteria of coeliac disease (CoD). At present it remains unclear whether they suffer from coeliac gluten sensitivity (CGS) or non-coeliac gluten sensitivity (NCGS). There are specific tissue markers of CoD such as anti-transglutaminase deposits (tTG) and intraepithelial lymphocytes expressing T-cell receptor (TCR) gamma/delta+.

Aim: To demonstrate the existence of CGS in these patients despite having negative celiac serology.

Methods: Double-blind randomized clinical trial of gluten vs placebo rechallenge for 6 months in patients with LE on a GFD. Inclusion criteria: >18 years, initial presentation with GI symptoms, HLA-DQ2/8+, negative celiac serology, good clinical and histological response to GFD. Patients were randomised to gluten (20 g/day) and placebo (maltrodextrin) (identical powder sachets mixed with meals). Clinical symptoms were analysed using visual analogue scales. Quality of life (GIQLI), adherence to diet, serology, and histological changes including gamma/delta+ IEL and tTG deposits were evaluated.

DETAILED DESCRIPTION:
Duodenal intraepithelial lymphocytosis (lymphocytic enteritis, LE) is defined by normal villous architecture and intraepithelial lymphocytes (IEL) >25/100 enterocytes. It is a frequent finding present in 2% to 5,4% of duodenal biopsies.

LE is secondary to coeliac disease (CoD) in only a minority of patients, since it may be a response to other inflammatory processes in the gut. Other possible aetiologies of LE include infections (Helicobacter Pylori), drugs (nonsteroidal anti-inflammatory or acetylsalicylic acid) and autoimmune disease. Observational studies have established CoD to account for 10% to 43% of cases with LD and positive HLA-DQ2/8 after undertaking an exhaustive diagnostic work-up. These 'minor' forms of CoD may have similar clinical manifestations to those with villous atrophy.

However, these patients with 'minor' CoD have often negative celiac serology, and then do not fulfil the present criteria to diagnose CoD. In fact, using the present diagnostic criteria they should be included in the definition of non-celiac gluten sensitivity (NCGS). For diagnosing NCGS it is necessary to rule out CoD by means of negative serology -endomysial and tissue transglutaminase IgA antibodies- and a duodenal biopsy with absence of villous atrophy on a gluten-containing diet. As such it is accepted that NCGS patients might have LE. A recent systematic review on NCGS revealed that 44% of patients presented HLA-DQ2/8 haplotypes, suggesting that a subgroup of patients with NCGS may actually belong in the spectrum of CoD, which some authors have so-called 'coeliac lite' disease.

The gold-standard assay for confirming NCGS requires dietary elimination, followed by double-blind, randomized, placebo-controlled food challenge. This procedure is difficult to adopt routinely in clinical practice. To date two double-blind placebo-controlled dietary interventions in patients with presumptive NCGS have been published. The first gluten vs placebo rechallenge trial showed that patients who received gluten had significantly more abdominal symptoms than those on placebo (68% vs 40%). The second study that investigated the specific effects of gluten after dietary reduction of fermentable, poorly absorbed, short-chain carbohydrates (FODMAPs) in subjects believed to have NCGS, showed no symptomatic worsening after gluten challenge as compared to placebo. Thus, there was no evidence of specific or dose dependent effect of gluten on NCGS patients placed on a diet low in FODMAPs. It is worth mentioning that patients included in these trials were HLA-DQ2/8 negative, and if positive they had a normal duodenal biopsy (Marsh 0) while on a gluten containing diet. Besides, a GFD has been shown to be more effective in IBS-D patients with negative CoD serology but HLA-DQ2/8+ than in those with a negative genetic study.

The recent ESPGHAN guidelines for CoD diagnosis suggest that in cases with low-grade enteropathy (including LE) both a high γδ IEL count and the presence of Ig A anti-tissue transglutaminase (anti-TG2) deposits in the mucosa increase the likelihood of CoD. In contrast to CoD, there is stated that in NCGS there is not an increase of T-cell receptor γδ IELs. However, these parameters have only been scarcely used to rule out CoD in patients with NCGS in literature.

The aim of study was demonstrate the existence of gluten sensitivity in patients with HLA-DQ2/8+, LE and negative celiac serology, who had presented a clinical and histological response to a gluten-free diet (GFD), using a gluten vs placebo-controlled challenge. In addition, to assess the presence of tissue markers of CoD before and after gluten challenge, thus confirming the existence of a 'coeliac-lite' disease.

ELIGIBILITY:
Inclusion Criteria:

1. Giving written informed consent
2. Patients with age ≥18 years
3. Histological diagnosis confirmed of lymphocytic enteritis (LE)
4. Celiac genetic study (HLA-DQ2 and /or HLA-DQ8 positive)
5. Negative serology of celiac disease
6. Previous complete clinical and histological response to gluten-free diet
7. Initial (at diagnosis) GI symptoms with or without extraintestinal manifestations.
8. No previous studies on both IEL cytometric pattern and anti-TG2 IgA subepithelial deposits.

Exclusion Criteria:

1. Patients who are unable to adhere to the study visit schedule and other protocol requirements according to the investigator.
2. Participation in a clinical trial in the last 30 days, simultaneous participation in a trial or prior participation in this study.
3. Previous diagnosis with gluten-sensitive enteropathy with villous atrophy and positive serology.
4. Patients with LE and initial response to gluten free diet but that at the time of inclusion are on a normal gluten-containing diet.
5. Severe co-morbidities.
6. Drug or alcohol abuse.
7. Pregnancy or breast-feeding.

At the initial diagnosis, other LE aetiologies, like non-steroidal anti-inflammatory drugs intake, parasitic infection, and Helicobacter pylori infection, were appropriately ruled out.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Clinical relapse | 6 months
  Visual analogue scale on clinical symptoms at each visit (Baseline, 4 weeks, 12 weeks, 24 weeks)

SECONDARY OUTCOMES:
Changes in health related quality of life | Change from baseline at 6 months (or premature withdrawn)
  GI quality of life index (GIQLI) at basal and 24 week visits
Histological evolution (Changes in intraepithelial lymphocyte count) | Changes from baseline at 6 months (or premature withdrawn)
  Changes in intraepithelial lymphocyte count
Changes in gamma/delta cells | Changes from baseline at 6 months (or premature withdrawn)
  Changes in cytometric count of gamma/delta cells
Changes in transglutaminase deposits | Changes from baseline at 6 months (or premature withdrawn)
  Presence of tTG deposits (IF)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fernández-Bañares, MD, Principal Investigator — Hospital Mutua Terrassa

REFERENCES:
- [Background] Molina-Infante J, Santolaria S, Sanders DS, Fernandez-Banares F. Systematic review: noncoeliac gluten sensitivity. Aliment Pharmacol Ther. 2015 May;41(9):807-20. doi: 10.1111/apt.13155. Epub 2015 Mar 6. PMID 25753138
- [Background] Fernandez-Banares F, Carrasco A, Garcia-Puig R, Rosinach M, Gonzalez C, Alsina M, Loras C, Salas A, Viver JM, Esteve M. Intestinal intraepithelial lymphocyte cytometric pattern is more accurate than subepithelial deposits of anti-tissue transglutaminase IgA for the diagnosis of celiac disease in lymphocytic enteritis. PLoS One. 2014 Jul 10;9(7):e101249. doi: 10.1371/journal.pone.0101249. eCollection 2014. PMID 25010214
- [Background] Rosinach M, Esteve M, Gonzalez C, Temino R, Marine M, Monzon H, Sainz E, Loras C, Espinos JC, Forne M, Viver JM, Salas A, Fernandez-Banares F. Lymphocytic duodenosis: aetiology and long-term response to specific treatment. Dig Liver Dis. 2012 Aug;44(8):643-8. doi: 10.1016/j.dld.2012.03.006. Epub 2012 Apr 11. PMID 22497904
- [Derived] Rosinach M, Fernandez-Banares F, Carrasco A, Ibarra M, Temino R, Salas A, Esteve M. Double-Blind Randomized Clinical Trial: Gluten versus Placebo Rechallenge in Patients with Lymphocytic Enteritis and Suspected Celiac Disease. PLoS One. 2016 Jul 8;11(7):e0157879. doi: 10.1371/journal.pone.0157879. eCollection 2016. PMID 27392045